CLINICAL TRIAL: NCT02867501
Title: Venous Distension in Patients With Aneurysmatic Arterial Disease Compared to the Venous Distension in Patients With Arterial Occlusive Disease
Brief Title: Venous Distension in Patients With Aneurysmatic Arterial Disease
Status: Completed | Type: Observational
Sponsor: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Principal Investigator, Janis Christian Bartelt, intern, Kantonsspital Baselland Bruderholz
Other Study IDs: 2016-00375
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Aortic Aneurysm, Abdominal; Popliteal Artery Aneurysm; Peripheral Arterial Occlusive Disease; Vascular Diseases; Aortic Diseases; Varicose Veins
Keywords: venous distension; venous reflux
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Popliteal Artery Aneurysm; Peripheral Arterial Occlusive Disease 1; Vascular Diseases; Aortic Diseases; Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Aneurysmatic disease: Patients with dilatative arteriopathy (DA) the aortic diameter must be > 3 cm or the popliteal artery diameter > 1.5 cm
- Peripheral arterial occlusive disease: Patients with arterial occlusive disease (PAOD) defined with an Ankle brachial index (ABI) < 0.9 and positive criteria in the Edinburgh questionnaire.
- Healthy: Control group of age matched persons without PAOD (ABI > 0.9) and without DA.

SUMMARY:
The aim of the study is to assess if venous distension in patients with aneurysmatic arteriopathy is higher compared to patients with peripheral arterial occlusive disease (PAOD) and in controls.

DETAILED DESCRIPTION:
Patients with aortic aneurysm and patients with PAOD and Controls will be investigated in the following manner: Duplexsonography with assessment of the arterial diameters in the aorta and leg arteries. Duplexsonography with assessment of venous reflux in proximal and deep veins of both legs Duplexsonography testing of venous distension in the common femoral vein, the great saphenous vein and the femoral vein.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dilatative arteriopathy (DA) the aortic diameter must be > 3 cm or the popliteal artery diameter > 1.5 cm
* Patients with arterial occlusive disease (PAOD) defined with an Ankle brachial index (ABI) < 0.9 and positive criteria in the Edinburgh questionnaire
* Patients able to give informed consent
* Control group of age matched persons without PAOD (ABI > 0.9) and without DA

Exclusion Criteria:

* Impossibility to stand
* Diabetes
* No given informed consent
* Persons and patients < 18 years old
* Acute deep venous thrombosis
* History of deep venous thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population is selected from patients of the angiologic clinic Baselland Bruderholz
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Venous distension of > 27% in patients with aneurysmatic arterial disease | one year

REFERENCES:
- [Background] Jeanneret C, Baldi T, Hailemariam S, Koella C, Gewaltig J, Biedermann BC. Selective loss of extracellular matrix proteins is linked to biophysical properties of varicose veins assessed by ultrasonography. Br J Surg. 2007 Apr;94(4):449-56. doi: 10.1002/bjs.5630. PMID 17262753
- [Background] Jeanneret C, Jager KA, Zaugg CE, Hoffmann U. Venous reflux and venous distensibility in varicose and healthy veins. Eur J Vasc Endovasc Surg. 2007 Aug;34(2):236-42. doi: 10.1016/j.ejvs.2007.03.018. Epub 2007 May 24. PMID 17524680